CLINICAL TRIAL: NCT05485259
Title: Effect of Alpha-lipoic Acid Supplementation on Regression of Low-grade Squamous Intraepithelial Lesions (LSIL)-Double Blind, Randomized, Placebo-controlled Trial
Brief Title: Effect of Alpha-lipoic Acid on Regression of Low-grade Squamous Intraepithelial Lesions (LSIL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: University Clinical Center Tuzla (Other)
Responsible Party: Principal Investigator, Dubravka Vitali Čepo, Prof., University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALA-SIL-1719
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Low-Grade Squamous Intraepithelial Lesions
Keywords: alpha-lipoic acid; low-grade squamous intraepithelial lesions; LSIL; CIN; cervical intraepithelial neoplasia.
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DL-alpha lipoic acid (Experimental): 600 mg (2x300 mg) of DL-alpha lipoic acid in capsules, per os daily for 3 months
  Interventions: Dietary Supplement: DL-alpha lipoic acid
- Placebo (Placebo Comparator): 600 mg (2*300 mg) of placebo (rice starch) in capsules, per os, daily for 3 months
  Interventions: Other: placebo (rice starch)

INTERVENTIONS:
Dietary Supplement: DL-alpha lipoic acid — Treatment group recieves 600 mg of DL-alpha lipoic acid daily, per os, for 3 months.
  Arms: DL-alpha lipoic acid
Other: placebo (rice starch) — Placebo group recieves 600 mg (2x300 mg) of placebo (rice starch) daily, per os, for 3 months
  Arms: Placebo

SUMMARY:
Low-grade squamous intraepithelial lesions (LSIL) are premalignant changes on the cervix that can lead to malignant changes, i. e. cervical cancer. Alpha-lipoic acid is a fatty acid that is naturally found in food, and due to its proven antioxidant and anti-inflammatory effects, it is increasingly used as a dietary supplement, most often to alleviate the symptoms of various neuropathic conditions.

The purpose of this study was to demonstrate efficiency, safety, and clinical benefit of alpha lipoic acid (ALA) in inducing regression of LSIL. The hypothesis is based on the proven role of oxidative stress and inflammation in formation of LSIL and anti-inflammatory and antioxidative efficiency of ALA.

The study was designed as randomized, double-blind, two-arm, placebo-control trial recruiting 100 female patients with diagnosed LSIL. Patients received 600 mg/day of ALA or placebo for 3 months. Progression/regression of LSIL has been defined as primary outcome of the study; inflammation markers and oxidative stress parameters have been defined as secondary outcomes of the study.

DETAILED DESCRIPTION:
Cervical intraepithelial neoplasia (CIN) is premalignant change on the cervix that can lead to malignant changes, i.e., cervical cancer. Today, this term has been replaced by the more recent term squamous intraepithelial lesion (SIL). With the introduction of the term SIL into use (as proposed by Bethesda system), two grades are used to classify premalignant changes of the cervix: SIL of low grade (LSIL) which includes condylomas and mild dysplasia (CIN I), and high-grade squamous intraepithelial lesion (HSIL) that includes changes in terms of medium and high-grade dysplasia (CIN II and CIN III). The main etiological factor that leads to the formation of cervical neoplasia is the human papilloma virus (HPV). Other etiological factors such as smoking, oral therapy contraceptives, sexual habits, chemicals, immunosuppressive therapy, immunodeficiency diseases, socioeconomic living conditions and nutritional status of patients also play a role in the progression of the disease. In addition to the above, inflammation and oxidative stress are also important etiological factors in the development of SIL. Namely, malignant changes on the cervix do not appear on a completely healthy cervix but are always associated with chronic cervicitis.

Alpha-lipoic acid (ALA) is a non-essential fatty acid with numerous metabolic roles and its therapeutic potential is being investigated in many pathophysiological conditions. In addition to acting as a cofactor of numerous signalling pathways in the cell, ALA also has a standard redox potential of -0.32 V, which gives it the ability to regenerate the most important physiological antioxidants in vivo (e.g. vitamin C and E) and makes it one of the most potent natural antioxidants. Given that it is implicated as a modulator of various inflammatory signalling pathways, its anti-inflammatory properties have been investigated by a large number of clinical studies. T This impressive array of cellular and molecular functions has led to significant interest in the research and use of ALA as a dietary supplement. ALA has been proven to improve insulin resistance, relieve symptoms of diabetic neuropathy, combine with phototherapy in the treatment of vitiligo, improve wound healing and increase the effectiveness of reduction diets. Its use as a dietary supplement is currently being investigated in dementia, burning mouth syndrome, carpal syndrome, glaucoma, cataracts, hypertension, and peripheral arterial disease. For therapeutic purposes, ALA is administered orally in doses of 300-1800 mg/day, and for some indications its topical and parenteral administration has been investigated. The safety of oral administration in the mentioned doses has been investigated in many clinical studies lasting from 4 months to 4 years. The effectiveness of ALA in premalignant changes of the cervix has not been investigated to date. Considering the proven effectiveness of oral supplementation with other antioxidants (such as green tea polyphenols or Se) in patients with LSIL, the aim of this research is to investigate, for the first time, the effectiveness of ALA in regression of LSIL.

The study was designed as double-blind, randomized, placebo-controlled trial where participants were asked to self-administer either 600 mg of ALA in form of 2 capsules containing 300 mg of ALA (donated by Zada Pharmaceuticals, Lukavac, Bosnia and Herzegovina) or a placebo (provided as identical oral capsules containing rice starch, also donated by Zada Pharmaceuticals) per os daily for 3 months. The research protocol for this study has been approved by the Ethics Committee of the University of Zagreb, Faculty of Pharmacy and Biochemistry and the Ethics Committee of the University Clinical Centre Tuzla. The trial was performed in accordance with the international, national, and institutional guidelines pertaining to clinical studies and biodiversity rights and it complied with the CONSORT guidelines.

At the initial appointment eligible patients were introduced to the study design. They were informed about the study protocol: aim and the purpose of the study, general methodology, expected roles of the participants, potential risks of participating in the study, potential benefits of the participation in the study, data confidentiality issues, and contact details of investigators who, when necessary, provided any kind of additionally needed information. In case patient agreed to participate in the study, they l signed informed consent form. All participants were asked to give their written informed consent for the inclusion in the study. After inclusion in the study patients filled a baseline questionnaire and provided information on basic anthropometric characteristics, reproductive history, current medication, and major lifestyle characteristics (smoking, level of physical activity). Examination of patients' eating and living habits was conducted using a standardized and validated semiquantitative food frequency questionnaire (FFQ) with the help of trained staff. Patients were advised not to change their diet during the study.

Participants were randomized in the ratio 1:1 for ALA: placebo. Patients were randomly allocated a patient number that determined their supplement allocation. They received two bottles of capsules prelabelled with their study number containing either capsules of ALA sufficient for 3 months of supplementation, or identical capsules of placebo (rice starch) sufficient for 3 months of supplementation. Patients were asked to return the remaining capsules after the 3-month period to assess the adherence. During the supplementation period participants were contacted twice by telephone by a research team member to check possible adverse effects and to improve the adherence. Compliance after enrolment was measured as the percentage of pills taken between visits. Subjects who took less than 75% of pills after randomization were considered as noncompliant and were taken off the study. 3 months after the entry participants were invited to a follow up appointment.

At both initial and follow-up appointment cytological screening, colposcopy and targeted biopsy and histological confirmation of cytological-colposcopic diagnosis wasconducted and blood samples were taken and analysed (assessment of primary and secondary outcomes of the study). The samples were collected at the Gynaecology and Obstetrics Clinic of the University Clinical Centre Tuzla over a period of 18 months. Sample analyses were conducted at the University Clinical Centre Tuzla and University of Zagreb, Faculty of Pharmacy and Biochemistry. Statistical processing, analysis and interpretation of the study results was completed within 6 months from the end of the analysis of the biological samples.

Patients' personal data, data on their lifestyle and eating habits (obtained from the FFQ) and measurements of the primary and secondary outcomes of the study were stored and processed in electronic form of the patients' registry. Data dictionary containing detailed descriptions of each variable used by the registry, including the source of the variable was developed. The registry was operated according to standard operative procedures of the University Clinical Centre Tuzla. Project manager and his associates were obliged to fully comply with the prescribed procedures for the protection of personal data. Patients' data were entered into project databases according to the initials of patients first and last name and using a special code. Their medical documentation was only reviewed by the project manager and his associates, and patients' name was never revealed to third parties. Patients' documentation was accessible to representatives of the Ethics Committee at the institution where clinical study was conducted (University Clinical Centre Tuzla) and representatives of the Committee for the Ethics of Experimental Work of the Faculty of Pharmacy and Biochemistry of the University of Zagreb, which is responsible for approving and supervising the conduct of this research.

Block randomization of patients was performed to ensure balance using an in-house computer program. To determine the sample size, a randomized clinical trial sample size formula was used, where type one (α) error was set at 5% and the study power was set at 90%. Ratio of case to control was 1, and expected dropout was 2%. LSIL wasthe main outcome of the study; expected proportion of LSIL in control group was 50%, and in the treated group 40%. Assuming a dropout 2% the target sample size has been determined to be 96 (48 subjects per group). The research results (qualification of cervical squamous epithelium lesions, parameters of inflammation, parameters of oxidative stress) was statistically processed using the MedCalc software package. The basic features of the variables were tested using descriptive analysis. The normality of data distribution was tested using the Kolmogorov-Smirnov test, and parametric or non-parametric statistical tests were used for further analysis of the results.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmation of a low degree of LSIL,
* sexually active women.

Exclusion Criteria:

* pregnancy
* malignant diseases
* diabetes
* chronic inflammatory diseases
* hysterectomy
* destructive therapy of the cervix
* abortion
* HPV vaccination
* menopause

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Regression of Low-Grade Squamous Intraepithelial Lesions (LSIL) | baseline to week 12
  LSIL will be confirmed by cytological screening, colposcopic examination of the cervix and targeted biopsy and histological confirmation of cytological-colposcopic diagnosis at the study baseline and after 3 months the intervention (day 0 and day 90). The findings of cytological screenings will be qualified according to the internationally recognized form "Zagreb 2002". The colposcopic form "Rio de Janeiro-Zagreb 2011" will be used to classify the colposcopic findings. Uterine tissue samples obtained by targeted colposcopic biopsy will be processed by a standard histological method. Assessment of the pathological diagnosis will be done as blindness by a single experienced pathologist at baseline and after the 3 months of intervention. The classification of premalignant and invasive cervical squamous epithelial lesions will be determined according to the WHO Tumour Classification.

SECONDARY OUTCOMES:
Change of oxidative stress parameters (serum antioxidant status) | baseline to week 12
  For the assessment of the secondary outcomes blood samples will be collected at baseline (day 0) and after the treatment (after 12 weeks) by venipuncture after a 10 h fasting period, aliqoted and stored at -20C for future analysis. Analyses will be conducted within 30 days from sample aquisition. The following oxidative stress parameters will be determined:
  total serum antioxidant status (assessed by measuring scavenging activity against the 2,2'-azino-bis(3-ethylbenzthiazoline-6-sulfonic acid radical (ABTS+˙); oxygen radical absorbance capacity (ORAC) of the serum and ferric reducing power of the serum (FRAP)); serum malondyaldehide levels (MDA); serum reduced glutathione levels (GSH); serum superoxide dismutaze activity (SOD).
Change of inflammation markers | baseline to week 12
  For the assessment of the secondary outcomes blood samples will be collected at baseline (day 0) and after the treatment (after 12 weeks) by venipuncture after a 10 h fasting period, aliqoted and stored at -20C for future analysis. Analyses will be conducted within 30 days from sample aquisition. The following inflammation parameters will be determined:
  fibrinogen; high-sensitive C-reactive protein; sedimentation; interleukin-6
Change of lipid parameters (lipoprotein profile) | baseline to week 12
  For the assessment of the secondary outcomes blood samples will be collected before and after the treatment at three months by venipuncture after a 10 h fasting period. Lipid parameters will be determined immediatelly after sample collection and include:
  measurement of triglycerides; measurement of total cholesterol; measurement of high-density lipoproteins (HDL ) measurement of low-density lipoproteins (LDL )

CONTACTS AND LOCATIONS:
Overall Officials: Dubravka Vitali Čepo, prof, Principal Investigator — University of Zagreb, Faculty of Pharmacy and Biochemistry; Zinaida Karasalihović, prof, Study Director — University Clinical Center Tuzla
Locations (2):
- University Clinical Center Tuzla, Tuzla, Bosnia and Herzegovina
- University of Zagreb, Zagreb, Dep. of Food Chemistry, Croatia

IPD SHARING:
Plan to Share IPD: No